CLINICAL TRIAL: NCT01871038
Title: A Case-Control Study to Assess the Effectiveness of Rotarix Vaccine (RV1)
Brief Title: Effectiveness of Monovalent Rotavirus Vaccine (RV1)
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: GlaxoSmithKline (Industry); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 111725
Record Dates: First submitted 2013-05-01; First posted 2013-06-06 (Estimated); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Rotavirus; Acute Gastroenteritis
Keywords: vaccine effectiveness; rotavirus; acute gastroenteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rotavirus Positive Cases: This group includes all participants who submitted a stool specimen that tested positive for Rotavirus.
- Rotavirus Negative Controls: This group includes all participants who submitted a stool specimen that tested negative for Rotavirus.

SUMMARY:
To determine the effectiveness of rotavirus vaccines, active surveillance will be conducted at two sites, Cincinnati Children's Hospital Medical Center (CCHMC) in Cincinnati, Ohio and the Medical University of South Carolina (MUSC) in Charleston, South Carolina.

Children born on or after April 1, 2006 presenting to CCHMC as an inpatient or for a short-stay or Emergency Department (ED) visit with acute gastroenteritis (AGE) and/or fever will be approached for enrollment. Children will be eligible if they have vomiting and/or diarrhea less than or equal to 10 days duration. Data including demographic information, illness characteristics and socio-economic status will be collected from each patient. A sample of the patient's stool will be collected within 14 days of the onset of symptoms. Stool specimens will be tested for rotavirus antigen by Rotaclone at CCHMC. All rotavirus positive stool specimens will be typed for common G and P serotypes. Using the children identified with rotavirus as our cases and the children who were rotavirus negative as our controls, we will conduct a case control study to assess the effectiveness of rotavirus vaccines, in particular Rotarix.

DETAILED DESCRIPTION:
A case-control design will be utilized to assess the effectiveness of RV1 in preventing rotavirus-associated hospitalizations and Emergency Department (ED) visits using cases and controls from the 2009-2012 rotavirus seasons. Vaccine exposure among cases will be compared to vaccine exposure among controls. There will be one case group and one control group.

Cases will be obtained from children who are enrolled in active surveillance for acute gastroenteritis being conducted at the two initial surveillance sites. These sites include: Cincinnati Children's Hospital Medical Center (2009-2012) and the Medical University of South Carolina (2009-2012). Cases and controls will be identified retrospectively for the 2008-2011 seasons and prospectively through active surveillance for the 2011-2012 season. The active surveillance programs conduct prospective surveillance for hospitalizations and ED visits due to AGE (acute gastroenteritis) in children < 6 years of age. Even though Rotarix was commercially available on January 1, 2008, the actual date that RV1 was initially used varied across sites. The date that Rotarix was initially used will be determined for each site through examination of the data. Children with laboratory-confirmed rotavirus infection (bulk stool sample positive for rotavirus using a rotavirus EIA) will be included as a case if they were born 2 months prior to the initial date of Rotarix availability at each site. The vaccine record for each case will be obtained to determine the vaccine status of the child.

Controls will be children born 2 months prior to the availability of Rotarix at each site who were enrolled in the active surveillance program at either site and who tested negative for rotavirus. Children who have been previously hospitalized for diarrhea, who have a sibling enrolled in the study, or who have recently moved into the study area (and might not have been eligible for the vaccine) will be excluded.

Laboratory Testing

For children enrolled in the active surveillance program bulk stool specimens are obtained within 14 days of the visit for AGE symptoms and are tested using Rotaclone, a commercial enzyme immunoassay (Meridian Bioscience, Inc) at CCHMC. Children with a positive test for rotavirus are eligible to be cases and children with a negative test for rotavirus are eligible for controls. Specimens positive by EIA for rotavirus will have G and P genotyping done at CCHMC.

Retrospective Enrollment of Children Tested for Rotavirus as Part of Routine Care

With the dramatic decline in rotavirus since the introduction of rotavirus vaccines, the number of children enrolled in surveillance has plummeted compared to pre-licensure surveillance. In order to improve our sample size, we will retrospectively invite children who had a rotavirus test done from August 1, 2008 through June 30, 2012 to participate in this study. The laboratory records of rotavirus testing will be reviewed to identify children with a date of birth >August 1, 2008. Once identified, a letter will be sent to the parents/guardians with a brief explanation of the study and we will ask them to notify us within two weeks if they do not wish to be called. Study staff will then contact the parent/guardian to explain the study and to determine whether the child meets eligibility criteria (same as those outlined for enrollment into surveillance). If the child meets eligibility criteria, the parents/guardians will be asked to allow their child to participate, informed consent will be obtained for the child. If agreed, the same data collected on prospectively enrolled children will be collected and permission will be obtained to contact the child's health care provider for the child's immunization records.

Eligibility

The date that Rotarix was initially used will be determined for each site. Children born 2 months prior to the initial date or later will be eligible to be a case or control for this study. If a child is enrolled more than once during the same season, the visit at which the child tested positive for rotavirus will be selected for inclusion; if the child tested negative at all visits, the child's final visit will be selected for inclusion.

Sample Size

Sample size calculations were done for varying degrees of vaccine efficacy and vaccine coverage. With a vaccine uptake of 20%, 68 cases would allow a detection of vaccine effectiveness of 80% assuming a two-sided test with a significance level of 0.05 and 80% power. If the vaccine uptake is 30% only 44 cases would be needed to detect a vaccine effectiveness of 80%.

One must take into consideration that both cases and controls may have incomplete immunization series. If there are a sufficient number of cases, one dose vaccine efficacy will also be examined.

Statistical Analysis

Analyses will be performed using SAS® (Version 9.2 Cary, NC). Demographic and risk factor variables will be examined. Continuous, parametric data will be presented as mean ± standard deviation (SD); continuous, non-parametric data will be presented as median (inter-quartile range). Categorical data will be presented as frequency (percentage) by category. Continuous, parametric data will be analyzed with ANOVA or Student's t-test. Categorical data will be analyzed with chi-square or Fisher's Exact Test as appropriate.

Logistic Regression will be used to estimate Vaccine Effectiveness (VE) and 95% confidence intervals (CIs) from the adjusted odds ratios (aORs) by using the formula VE = (1-aOR) X 100. Cases and controls will be matched on age, enrollment date, and geographic region. Cases will be compared to matched controls in order to evaluate the effectiveness of full (2 doses) and partial (1 dose) vaccination. Initially, univariate conditional logistic regression analyses will be performed to determine which covariates should be included in the multivariable analysis. The explanatory variable of interest is vaccination status. If sample size permits, vaccine effectiveness will be calculated by serotype. Other possible covariates to be included are: date of birth, age at onset, season, insurance status (public/none versus private) and point of care (hospital or ED). Variables with p-values ≤ 0.20 will selected as candidates for multivariable analysis. Multicollinearity among the covariates will be examined by evaluating variance inflation factors. If collinearity is present, only one of the correlated variables will be entered into the model at a time. Analysis will be rerun choosing alternative correlated variables and the models will be compared. The model with the lowest Akaike information criterion (AIC) will be chosen as the final model. Model selection will include stepwise, forward selection, and backwards elimination. The Hosmer-Lemeshow test will be used to determine goodness of fit.

ELIGIBILITY:
Inclusion Criteria:

* the child is < 6 years of age
* for the vaccine effectiveness analysis using the Minimum Age Model, the child was included if born on or after 8/10/2008 at MUSC and on or after 12/1/2008 at CCHMC.
* for the vaccine effectiveness analysis using the Maximum Age Model, the child was included if >=8 months of age.
* the child is being evaluated at Cincinnati Children's Hospital Medical Center (CCHMC) or the Medical University of South Carolina (MUSC) as an inpatient, short-stay visit or in the emergency department
* the child has acute gastroenteritis defined as

  * diarrhea (>3 loose stools in a 24 hour period) OR
* -vomiting (>1 episodes in a 24 hour period)
* the child's illness is of <10 days duration
* written consent is obtained from the child's parent or legal guardian

Exclusion Criteria:

* the child is >6 year of age
* the child had onset of fever or gastroenteritis symptoms > 10 days prior to admission
* the child has a non-infectious or other identifiable cause of their symptoms, such as head trauma, pyelonephritis, pyloric stenosis, or prolonged coughing
* the child is immunocompromised
* there is no parent or guardian available
* the parent/guardian is non-English speaking
* previously enrolled for the same episode of gastroenteritis
* for the vaccine effectiveness analysis using the Minimum Age Model, the child was excluded if born prior to 8/10/2008 at MUSC and prior to 12/1/2008 at CCHMC.
* for the vaccine effectiveness analysis using the Maximum Age Model, the child was excluded if <8 months of age.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who are an inpatient or a patient of the Emergency Department with symptoms of acute gastroenteritis.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Staat, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children less than 6 years of age with hospitalizations and emergency department (ED visits due to AGE between 1/1/2008-6/30/2012 were prospectively recruited to participate in the study at Cincinnati Children's Hospital Medical Center (CCHMC) and the Medical University of South Carolina (MUSC).
Pre-assignment Details: 362 participants were enrolled in the overall study, which is stated in the protocol section. The participant totals in Models One and Two do not equal the overall number enrolled because some participants were included in both models.
Groups:
- Vaccine Effectiveness Study Population - Rotavirus Positive Cases: Patients eligible for active surveillance based on the recruitment details and eligibility criteria who provided a stool specimen to be tested that had a positive stool sample.
- Vaccine Effectiveness Study Population - Rotavirus Negative Controls: Patients eligible for active surveillance based on the recruitment details and eligibility criteria who provided a stool specimen to be tested that had a Negative stool sample.
Period: Overall Study
Arm/Group | Vaccine Effectiveness Study Population - Rotavirus Positive Cases | Vaccine Effectiveness Study Population - Rotavirus Negative Controls
Started | 49 | 313
Completed | 49 | 313
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were included in the parent provided informed consent, if an adequate stool specimen was provided, the child was <6 years of age, had symptoms <10 days duration that were consistent with acute gastroenteritis.
Groups:
- Rotavirus Positive Cases: All stool specimens were tested for rotavirus. Participants with a positive test result are included in this category.
- Rotavirus Negative Controls: All stool specimens were tested for rotavirus. Participants with a negative test result are included in this category.
- Total: Total of all reporting groups
Arm/Group | Rotavirus Positive Cases | Rotavirus Negative Controls | Total
Number analyzed (Participants) | 49 | 313 | 362
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 313 | 362
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: months] | 16.13 [2.1 to 35.7] | 14.82 [3.1 to 43.3] | 14.83 [2.1 to 43.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 149 | 167
  Male | 31 | 164 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 19 | 21
  Not Hispanic or Latino | 47 | 293 | 340
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 164 | 188
  White | 20 | 110 | 130
  More than one race | 4 | 26 | 30
  Unknown or Not Reported | 1 | 11 | 12
Region of Enrollment [Number; unit: participants]
  United States | 49 | 313 | 362
Vaccination Status [Count of Participants; unit: Participants] — Vaccination status:
  Partially vaccinated equal to single dose. Fully vaccinated equal to two doses.
  Participants
    Fully Vaccinated with Rotarix only | 12 | 193 | 205
    Partially Vaccinated with Rotarix only | 6 | 31 | 37
    Not Vaccinated | 31 | 89 | 120

OUTCOME MEASURES:

1. Primary Outcome: Matched VE Participants in the Minimum Age Model
Description: RV1 Vaccine Effectiveness (VE) was studied using a subset of the active surveillance participants who were at least 52 days of age. The recommend age for the first dose is 42 days, but children are considered vaccinated if they receive that dose within 4 days of the recommended age, which lowers the acceptable minimum age to 38 days. We added 14 days to enable them to mount an immune response to arrive at a minimum age of 52 days. We estimated RV1 VE of 2 doses vs 0 doses and 1 dose vs 0 doses.
Time Frame: 14 days from the date of enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Minimum Age Model - Rotavirus Positive Cases: All stool samples were tested using Rotaclone, a commercially available immunoassay and this group contain those participants that tested positive for rotavirus.
- Minimum Age Model - Rotavirus Negative Controls: All stool samples were tested using Rotaclone, a commercially available immunoassay and this group contain those participants that tested negative for rotavirus.
Arm/Group | Minimum Age Model - Rotavirus Positive Cases | Minimum Age Model - Rotavirus Negative Controls
Number analyzed (Participants) | 49 | 182
Participants
  O Doses | 31 | 70
  1 Dose | 6 | 31
  2 Doses | 12 | 81

2. Primary Outcome: Vaccine Effectiveness of RV1 in the Minmum Age Model
Description: RV1 Vaccine Effectiveness (VE) was studied using a subset of the active surveillance participants who were age-eligible to receive at least the first dose of RV1 vaccine. Only valid RV1 vaccinations were considered. We estimated RV1 VE of 2 doses vs 0 doses and 1 dose vs 0 doses. VE was estimated as (1 - exposure odds ratio) x 100.
Time Frame: 14 days from the date of enrollment
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- 2 vs 0 Doses in Minimum Age Model: We compared RV1 VE between participants that received 2 doses versus 0 doses of RV1.
- 1 vs 0 Doses in Minimum Age Model: We compared RV1 VE between participants what received 1 dose vs 0 doses of RV1.
Arm/Group | 2 vs 0 Doses in Minimum Age Model | 1 vs 0 Doses in Minimum Age Model
Number analyzed (Participants) | 194 | 138
percent probability | 69 [32 to 86] | 59 [-13 to 85]
Statistical Analysis 1: Comparison: 2 vs 0 Doses in Minimum Age Model; Test type: Superiority or Other; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.14 to 0.68] — Conditional logistic regression was used for matched analyses. Adjusted VE = (1 - adjusted OR) * 100
Statistical Analysis 2: Comparison: 1 vs 0 Doses in Minimum Age Model; Test type: Superiority or Other; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.15 to 1.13] — Conditional logistic regression was used for matched analyses. Adjusted VE = (1 - adjusted OR) * 100

3. Primary Outcome: Matched VE Participants in the Maximum Age Model
Description: RV1 Vaccine Effectiveness (VE) was studied using a subset of the active surveillance participants who were at least 8 months of age, the maximum recommend age for completion of 2 doses of RV1. We estimated RV1 VE of 2 doses vs 0 doses and 1 dose vs 0 doses.
Time Frame: 14 days from the date of enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Maximum Age Model - Rotavirus Positive Cases: All stool samples were tested using Rotaclone, a commercially available immunoassay and this group contain those participants that tested positive for rotavirus.
- Maximum Age Model - Rotavirus Negative Controls: All stool samples were tested using Rotaclone, a commercially available immunoassay and this group contain those participants that tested negative for rotavirus.
Arm/Group | Maximum Age Model - Rotavirus Positive Cases | Maximum Age Model - Rotavirus Negative Controls
Number analyzed (Participants) | 38 | 283
Participants
  0 Doses | 24 | 83
  1 Dose | 3 | 29
  2 Doses | 11 | 171

4. Primary Outcome: Vaccine Effectiveness of RV1 in the Maximum Age Model
Description: RV1 Vaccine Effectiveness (VE) was studied using a subset of the active surveillance participants who were greater than or equal to 8 months of age, the maximum recommended age for completion of two doses of RV1 vaccine. Only valid RV1 vaccinations were considered. We estimated RV1 VE of 2 doses vs 0 doses and 1 dose vs 0 doses. VE was estimated as (1 - exposure odds ratio) x 100.
Time Frame: 14 days from the date of enrollment
Measure: Number (95% Confidence Interval); unit: percentage probability
Groups:
- 2 vs 0 Doses in Maximum Age Model: We compared RV1 VE between participants that received 2 doses versus 0 doses of RV1.
- 1 vs 0 Doses in Maximum Age Model: We compared RV1 VE between participants what received 1 dose vs 0 doses of RV1.
Arm/Group | 2 vs 0 Doses in Maximum Age Model | 1 vs 0 Doses in Maximum Age Model
Number analyzed (Participants) | 289 | 139
percentage probability | 82 [59 to 92] | 77 [13 to 94]
Statistical Analysis 1: Comparison: 2 vs 0 Doses in Maximum Age Model; Test type: Superiority or Other; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.08 to 0.41] — Multivariable logistic regression including month and year of birth and month and year of symptom onset as covariates was used for unmatched analyses. Adjusted VE = (1 - adjusted OR) * 100
Statistical Analysis 2: Comparison: 1 vs 0 Doses in Maximum Age Model; Test type: Superiority or Other; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.06 to 0.87] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: From date of enrollment until sample collection, a maximum of 14 days.
Groups:
- Rotavirus Positive Cases: Cases are those participants who tested positive for rotavirus.
- Rotavirus Negative Controls: Controls are those participants who tested negative for rotavirus.
Arm/Group | Rotavirus Positive Cases | Rotavirus Negative Controls
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/313
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/313
Other Adverse Events (participants affected / at risk) | 0/49 | 0/313

LIMITATIONS AND CAVEATS:
Limitations of the study include very low numbers of rotavirus cases and temporary halt in use of Rotarix vaccine due to presence of porcine virus in the vaccine which resulted in several children receiving mixed doses of vaccine and a delayed uptake in Rotarix vaccine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No